CLINICAL TRIAL: NCT00771745
Title: Prospective, Single Center, Pilot Study of Pretransplant Thymoglobulin Administration and Early Corticosteroid Withdrawal in Living Donor Renal Transplant Recipients Under Mycophenolate Mofetil (MMF) and Tacrolimus Immunosuppression
Brief Title: Prospective Pilot Study of Pre-Transplant Thymoglobulin Administration in Living Donor Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, E. Steve Woodle, MD, FACS, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pre-Tx Thymo
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Renal Transplant Rejection; Transplants and Implants
MeSH Terms: interventions — thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rATG 4 doses (Active Comparator): Preloading Induction with Thymoglobulin® X 4 doses given day -4, day -2, day 0, and day 2 at 1.5 mg/kg/dose + corticosteroid taper + tacrolimus + MMF
  Interventions: Drug: Thymoglobulin
- rATG 3 doses (Active Comparator): Preloading Induction with Thymoglobulin® X 3 doses given day -4 (1.5mg/kg), day -2 (1.5mg/kg), and day 0 (3mg/kg) + corticosteroid taper + tacrolimus + MMF
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin — Preloading Induction with Thymoglobulin® X 4 doses given day -4, day -2, day 0, and day 2 at 1.5 mg/kg/dose + corticosteroid taper + tacrolimus + MMF
  Other Names: Anti-thymocyte globulin (rabbit), thymoglobulin; rATG
  Arms: rATG 4 doses
Drug: Thymoglobulin — Preloading Induction with Thymoglobulin® X 3 doses given day -4 (1.5mg/kg), day -2 (1.5mg/kg), and day 0 (3mg/kg) + corticosteroid taper + tacrolimus + MMF
  Other Names: anti-thymocyte globulin (rabbit), thymoglobulin; rATG
  Arms: rATG 3 doses

SUMMARY:
To determine how safe and effective giving Thymoglobulin before transplantation to patients who are going to be receiving kidney transplants.

DETAILED DESCRIPTION:
We will evaluate the therapeutic efficacy of administering Thymoglobulin® induction pre-transplantation in renal allograft recipients. Patients receiving pre-transplant Thymoglobulin will be evaluated for acute rejection (Banff '97 criteria), survival, and safety at 6 months. Overall the use of Thymoglobulin induction pre-transplantation will be safe and effective.

ELIGIBILITY:
Inclusion Criteria:

1. Adult living donor renal transplant recipient.
2. Patient is at least 18 years of age
3. If female and of childbearing potential, have a negative serum or urine HCG within 24 hours prior to Study Day -5 (Day of 1st Thymoglobulin dose) and must practice a medically approved method of birth control for the past 30 days prior to enrollment and agree to continue this practice during the 6 month efficacy analysis.
4. Signed informed consent.

Exclusion Criteria:

1. Human Leukocyte Antibody (HLA) identical living donor transplant recipient.
2. History of a positive cross-match with the donor.
3. Patients with a peak CDC PRA > 50% or a current CDC PRA > 25%.
4. Patients who have previously received a kidney transplant.
5. Active donor or recipient serology positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
6. History of noncompliance.
7. History of chronic corticosteroid or immunosuppressive use except for inhaled corticosteroids to treat asthma. .
8. Multiple organ transplant recipient.
9. Patient with a urinary bladder that is absent or not functional (e.g. self catheterization) pretransplant.
10. Patient who does not agree to use effective birth control during the 6-month efficacy analysis.
11. Known contraindication to administration of rabbit antithymocyte globulin.
12. Initial screening laboratory evaluations will be done locally before renal transplantation and the following laboratory values will be exclusionary: Platelets < 100,000/mm23 or WBC < 3000/mm3
13. Currently abusing drugs or alcohol or, in the opinion of the investigator, is at high risk for poor compliance.
14. Patient who, in the opinion of the investigator, has significant medical or psychosocial problems or unstable disease states that would preclude participation in the study. Examples of significant problems include, but are not limited to, morbid obesity or severe cardiac disease.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Steve Woodle, MD, Principal Investigator — University of Cincinnati; Adele Rike, PharmD, Principal Investigator — The Christ Hospital
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Preloading Induction With Thymoglobulin: Preloading Induction with Thymoglobulin® X 4 doses given day -4, day -2, day 0, and day 2 at 1.5 mg/kg/dose + corticosteroid taper + tacrolimus + MMF
  anti-thymocyte globulin (rabbit) : Preloading Induction with Thymoglobulin® X 4 doses given day -4, day -2, day 0, and day 2 at 1.5 mg/kg/dose + corticosteroid taper + tacrolimus + MMF
- Preloading Induction With Thymoglobulin® X 3 Doses: Preloading Induction with Thymoglobulin® X 3 doses given day -4 (1.5mg/kg), day -2 (1.5mg/kg), and day 0 (3mg/kg) + corticosteroid taper + tacrolimus + MMF
  anti-thymocyte globulin (rabbit) : Preloading Induction with Thymoglobulin® X 3 doses given day -4 (1.5mg/kg), day -2 (1.5mg/kg), and day 0 (3mg/kg) + corticosteroid taper + tacrolimus + MMF
Period: Overall Study
Arm/Group | Preloading Induction With Thymoglobulin | Preloading Induction With Thymoglobulin® X 3 Doses
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preloading Induction With Thymoglobulin | Preloading Induction With Thymoglobulin® X 3 Doses | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (17.1) | 36.1 (12.5) | 43.1 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Composite End Point of Acute Rejection, Graft Loss or Patient Death
Description: Proportion of Patients Meeting the Composite End Point of Acute Rejection, Graft loss or Patient death
Time Frame: 6 months
Population: Patients received tacrolimus (goal level 10-15 ng/mL) and mycophenolate mofetil (2gm daily) at time of transplant. Methylprednisolone (MP), acetaminophen, and diphenhydramine were given as premedication for each rATG dose (500mg MP 1st dose, 250mg MP subsequent 2 doses, 125mg MP 4th dose).
Measure: Number; unit: participants
Groups:
- Preloading Induction With Thymoglobulin x 4 Doses: Preloading Induction with Thymoglobulin® X 4 doses given day -4, day -2, day 0, and day 2 at 1.5 mg/kg/dose + corticosteroid taper + tacrolimus + MMF
  anti-thymocyte globulin (rabbit) : Preloading Induction with Thymoglobulin® X 4 doses given day -4, day -2, day 0, and day 2 at 1.5 mg/kg/dose + corticosteroid taper + tacrolimus + MMF
Arm/Group | Preloading Induction With Thymoglobulin x 4 Doses | Preloading Induction With Thymoglobulin® X 3 Doses
Number analyzed (Participants) | 6 | 5
participants
  Acute rejection | 1 | 1
  Patient Death | 0 | 0
  Graft Loss | 0 | 0

2. Secondary Outcome: Incidence of Treatment Failures: Defined as the Percentage of Patients That do Not Remain on Initial Therapy.
Time Frame: Ongoing
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Infections
Time Frame: Not defined
Reporting Status: Not Posted

4. Secondary Outcome: Need for Antilymphocyte Antibody Therapy to Treat Acute Rejection
Time Frame: Not defined
Reporting Status: Not Posted

5. Secondary Outcome: Severity of Biopsy-proven Rejection Using Banff 97 Criteria
Time Frame: Not defined
Reporting Status: Not Posted

6. Secondary Outcome: Serum Creatinine
Time Frame: Post-operative days 1-7, 30, 90 and 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Malignancy
Time Frame: Undefined
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Preloading Induction With Thymoglobulin | Preloading Induction With Thymoglobulin® X 3 Doses
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/5
Other Adverse Events (participants affected / at risk) | 4/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preloading Induction With Thymoglobulin (N=6) | Preloading Induction With Thymoglobulin® X 3 Doses (N=5)
Banff 1A Rejection (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient was admitted for acute renal failure. Biopsy showed Banff 1A rejection. Patient treated with solumedrol and IVIG.
Renal Allograft Dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient was admitted for renal allograft dysfunction. Biopsy was negative for rejection.
Acute Renal Failure / Anemia (Renal and urinary disorders) | 0 (0) | 1 (2) — Patient was admitted for acute renal failure and anemia. Biopsy was negative for rejection. Anemia was treated with Aranesp
Fever/Acute Renal Failure/Acidosis (Renal and urinary disorders) | 0 (0) | 1 (3) — Patient was admitted for fever of unclear etiology, acute renal failure and acidosis. Biopsy was negative for rejection. Patient treated with IV fluids for acidso
Increased Serum Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1) — Patient was admitted for a kidney biopsy due to a bump in her scr. Preliminary biopsy report shows diffuse inflammation, diffuse C4d positivity, humoral and cellular rejection with possible superimposed pyelonephritis.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preloading Induction With Thymoglobulin (N=6) | Preloading Induction With Thymoglobulin® X 3 Doses (N=5)
Fever / Chills (Immune system disorders) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Fever > 102°F (Immune system disorders) | 1 (1) | 1 (1)
Body Aches (General disorders) | 1 (1) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
PLT < 100,000 cells/mm3 (Investigations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No